CLINICAL TRIAL: NCT04037514
Title: Paracetamol Versus Ibuprofen in Premature Infants With Hemodynamically Significant Patent Ductus Arteriosus: a Randomized Clinical Trial
Brief Title: Paracetamol Versus Ibuprofen in Premature Infants With Hemodynamically Significant Patent Ductus Arteriosus
Acronym: IBUPAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Máximo Vento Torres (Other)
Collaborators: Instituto de Investigacion Sanitaria La Fe (Other); Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Sponsor-Investigator, Máximo Vento Torres, Scientific Director Health Research Institute La Fe, Instituto de Investigacion Sanitaria La Fe
Organization: Instituto de Investigacion Sanitaria La Fe (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IBUPAR-TRIAL
Record Dates: First submitted 2019-07-23; First posted 2019-07-30 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Patent Ductus Arteriosus After Premature Birth
MeSH Terms: interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paracetamol (Experimental): Intravenous paracetamol 15 mg/kg/6h for 3 or 6 days
  Interventions: Drug: Paracetamol
- Ibuprofen (Active Comparator): Intravenous ibuprofen 10 mg/kg/24 h (day 1) and 5 mg/kg/24h (day 2 and 3) for 3 or 6 days
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Paracetamol — Intravenous paracetamol 15 mg/kg/6h
  Arms: Paracetamol
Drug: Ibuprofen — Intravenous ibuprofen 10 mg/kg/24h (day 1) and 5 mg/kg/24h (day 2 and 3)
  Arms: Ibuprofen

SUMMARY:
Multicentric, double-blind clinical trial, which will evaluate the efficacy of iv paracetamol versus standard treatment with ibuprofen in the closure of patent ductus arteriosus in the preterm newborn. Secondarily, we intend to compare the safety of both treatments, increase our knowledge about the pharmacokinetics, pharmacodynamics and pharmacogenetics of paracetamol and ibuprofen in the neonatal period and make a pharmacoeconomic assessment of the use of both drugs.

DETAILED DESCRIPTION:
Those newborns ≤ 30 weeks of gestational age who are diagnosed in the first 2 weeks of hemodynamically significant ductus arteriosus and who do not meet any exclusion criteria will be eligible to participate in the study.

The PARACETAMOL group will receive intravenous doses of 15 mg/kg administered every 6h for 3 days (up to a maximum of 2 courses, i.e. 6 days). The IBUPROFEN group (control group) will receive the usual treatment, this is an initial dose of 10 mg/kg followed by 5 mg/kg intravenously at 24 and 48 hours after the first (all three doses are considered a treatment course), up a maximum of 2 courses).

A daily echocardiographic control will be performed to evaluate the closure of the ductus. If the ductus remains open and with significant clinical repercussion after completing a 3-day course of treatment, another batch of 3 doses of the same treatment will be administered. If medical treatment fails after two courses (6 days), the possibility of administering a batch of Ibuprofen at usual doses in both groups with the intention of offering standard treatment to all patients will be considered. Once the medical treatment with both drugs is completed if the ductus remains significant, the surgical closure will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed consent of parents/guardians
* Gestacional Age ≤30 weeks
* Postnatal age ≤ 2 weeks
* Need for ventilatory support
* Born in participating hospital/arrival to them within the period of application of the treatment
* 1 st episode of hemodynamically significant Patent Ductus Arteriosus

Exclusion Criteria:

* Major congenital malformations or chromosomopathies
* Refusal to participate and / or sign the informed consent.
* Impossibility or erroneous randomization
* Participation in another clinical trial with drugs
* Diuresis less than 1 ml / kg / h for 8 h prior to treatment
* Greater than 1.8 mg / dl Creatinine
* Platelets below 50,000 / uL
* Active bleeding (tracheal, gastrointestinal and renal)
* Intraventricular hemorrhage recently (48h) (grades 3-4)
* Severe hyperbilirubinemia
* Liver failure or severe coagulopathy
* Active necrotizing enterocolitis or intestinal perforation
* Septic shock
* Imminent death

Max Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 133 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Rate of closure of the hsPDA after treatment with paracetamol (experimental drug) versus ibuprofen (control drug). | 24-48 hours after the completion of study intervention
  It will include the closure rate after the first course of treatment, considered as ductus diameter < 1 mm monitored by echocardiography performed by a pediatric cardiology specialist.

SECONDARY OUTCOMES:
Need for a second course of treatment | from randomization until discharge, an average of 2 months
Closure rate after two treatment courses | from randomization until discharge, an average of 2 months
Need for rescue treatment after two courses of treatment | from randomization until discharge, an average of 2 months
Reopening rate after closure | from randomization until discharge, an average of 2 months
Closing rate after reopening | from randomization until discharge, an average of 2 months
Time required until closing | from randomization until discharge, an average of 2 months
Need for surgical ligation | from randomization until discharge, an average of 2 months
Incidence of early complications | from randomization until discharge, an average of 2 months
  oliguria, renal failure, necrotizing enterocolitis, intraventricular hemorrhage, hyperbilirubinemia, gastrointestinal bleeding or perforation
Incidence of late complications | from randomization until 2 years
  bronchopulmonary dysplasia, periventricular leukomalacia, necrotizing enterocolitis, retinopathy of the newborn, neurodevelopmental assessment, sepsis, death
Pharmacodynamics model of paracetamol in the context of hsPDA: Maximum Plasma Concentration [Cmax] | 24-48 hours after the completion of study intervention
  Relation of effectiveness/adverse reactions to serum levels
Pharmacodynamics model of paracetamol in the context of hsPDA: Minimum Plasma Concentration [Cmin] | 24-48 hours after the completion of study intervention
  Relation of effectiveness/adverse reactions to serum levels
Pharmacodynamics model of paracetamol in the context of hsPDA: Area Under the Curve [AUC]) | 24-48 hours after the completion of study intervention
  Relation of effectiveness/adverse reactions to serum levels
Pharmacodynamics model of paracetamol in the context of hsPDA: urine metabolites | 24-48 hours after the completion of study intervention
  Quantification of metabolites in urine and its relationship with drug elimination/metabolism
Pharmacogenetics of paracetamol | 24-48 hours after the completion of study intervention
  Genetic polymorphisms in TFAP2B, TGFBR2, EPAS1, MD-2 and GM2A genes related to efficacy/occurrence of adverse reactions
Price-effectiveness ratio. Cost-effectiveness analysis depending on the efficiency obtained in the treatment. | from randomization until discharge, an average of 2 months
Genotoxicity mesured by %DNA damage | from randomization until discharge, an average of 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Maximo Vento Torres, PhD, MD, Study Chair — Hospital Universitario La Fe
Locations (4):
- Spain (4):
  - Hospital Reina Sofía, Córdoba, Cordoba
  - Hospital Universitario de Cabueñes, Gijón, Gijón
  - Hospital Materno-Infantil (Hospital Regional Carlos Haya) Málaga:, Málaga, Málaga
  - Hospital Universitari i Politècnic La Fe, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dang D, Wang D, Zhang C, Zhou W, Zhou Q, Wu H. Comparison of oral paracetamol versus ibuprofen in premature infants with patent ductus arteriosus: a randomized controlled trial. PLoS One. 2013 Nov 4;8(11):e77888. doi: 10.1371/journal.pone.0077888. eCollection 2013. PMID 24223740
- [Background] Hammerman C, Bin-Nun A, Markovitch E, Schimmel MS, Kaplan M, Fink D. Ductal closure with paracetamol: a surprising new approach to patent ductus arteriosus treatment. Pediatrics. 2011 Dec;128(6):e1618-21. doi: 10.1542/peds.2011-0359. Epub 2011 Nov 7. PMID 22065264
- [Background] Oncel MY, Yurttutan S, Erdeve O, Uras N, Altug N, Oguz SS, Canpolat FE, Dilmen U. Oral paracetamol versus oral ibuprofen in the management of patent ductus arteriosus in preterm infants: a randomized controlled trial. J Pediatr. 2014 Mar;164(3):510-4.e1. doi: 10.1016/j.jpeds.2013.11.008. Epub 2013 Dec 18. PMID 24359938
- [Background] Yang B, Gao X, Ren Y, Wang Y, Zhang Q. Oral paracetamol vs. oral ibuprofen in the treatment of symptomatic patent ductus arteriosus in premature infants: A randomized controlled trial. Exp Ther Med. 2016 Oct;12(4):2531-2536. doi: 10.3892/etm.2016.3676. Epub 2016 Sep 6. PMID 27698754
- [Background] Dash SK, Kabra NS, Avasthi BS, Sharma SR, Padhi P, Ahmed J. Enteral paracetamol or Intravenous Indomethacin for Closure of Patent Ductus Arteriosus in Preterm Neonates: A Randomized Controlled Trial. Indian Pediatr. 2015 Jul;52(7):573-8. doi: 10.1007/s13312-015-0677-z. PMID 26244949
- [Background] Sancak S, Gokmen Yildirim T, Topcuoglu S, Yavuz T, Karatekin G, Ovali F. Oral versus intravenous paracetamol: which is better in closure of patent ductus arteriosus in very low birth weight infants? J Matern Fetal Neonatal Med. 2016;29(1):135-9. doi: 10.3109/14767058.2014.989829. Epub 2014 Dec 23. PMID 25471090
- [Background] El-Khuffash A, Jain A, Corcoran D, Shah PS, Hooper CW, Brown N, Poole SD, Shelton EL, Milne GL, Reese J, McNamara PJ. Efficacy of paracetamol on patent ductus arteriosus closure may be dose dependent: evidence from human and murine studies. Pediatr Res. 2014 Sep;76(3):238-44. doi: 10.1038/pr.2014.82. Epub 2014 Jun 18. PMID 24941212
- [Derived] Garcia-Robles A, Gimeno Navarro A, Serrano Martin MDM, Parraga Quiles MJ, Parra Llorca A, Poveda-Andres JL, Vento Torres M, Aguar Carrascosa M. Paracetamol vs. Ibuprofen in Preterm Infants With Hemodynamically Significant Patent Ductus Arteriosus: A Non-inferiority Randomized Clinical Trial Protocol. Front Pediatr. 2020 Jul 17;8:372. doi: 10.3389/fped.2020.00372. eCollection 2020. PMID 32766181